CLINICAL TRIAL: NCT06109649
Title: A Double-Arm, Open Label, Phase III Study to Compare the Efficacy and Safety of SCENESSE and Narrow-Band Ultraviolet B (NB-UVB) Light Versus NB-UVB Light Alone in the Treatment of Vitiligo
Brief Title: A Study to Compare the Efficacy and Safety of SCENESSE and Narrow-Band Ultraviolet (NB-UVB) Light Versus NB-UVB Light Alone in Patients With Vitiligo
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Clinuvel, Inc. (Industry)
Responsible Party: Sponsor
Organization: Clinuvel Pharmaceuticals Limited (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUV105
Record Dates: First submitted 2023-10-20; First posted 2023-10-31 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-02

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — afamelanotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Afamelanotide and NB-UVB Light (Experimental)
  Interventions: Drug: Afamelanotide and NB-UVB Light
- NB-UVB Light (Other)
  Interventions: Procedure: NB-UVB Light

INTERVENTIONS:
Drug: Afamelanotide and NB-UVB Light — Patients will receive combination of NB-UVB twice weekly and afamelanotide every 3 weeks for 20 weeks.
  Arms: Afamelanotide and NB-UVB Light
Procedure: NB-UVB Light — Patients will receive NB-UVB light twice per week for 20 weeks. Upon study completion, NB-UVB Light Arm participants will have the opportunity to enroll in an open-label extension phase of the study. In this extension phase, participants will undergo the same evaluations and assessments as the ones performed in the main part of the study under Afamelanotide and NB-UVB Light Arm.
  Arms: NB-UVB Light

SUMMARY:
The CUV105 study will assess the efficacy and safety of afamelanotide and NB-UVB light in patients with vitiligo on the body and face versus NB-UVB light alone.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with a confirmed diagnosis of generalized vitiligo with VASI≥3 of the body and VASI on the head and neck ≥0.3 including an F-VASI≥0.1
* Stable or active vitiligo
* Aged 12 or more
* Fitzpatrick skin types III-VI

Exclusion Criteria:

* Fitzpatrick skin types I-II
* Extensive leukotrichia
* Treatment with NB-UVB phototherapy in the last three months prior to study start
* Allergy to afamelanotide or the polymer contained in the implant
* Any other treatment for vitiligo within 30 days prior to the Screening Visit
* History of melanoma or lentigo maligna
* History of dysplastic nevus syndrome
* Any malignant skin lesions
* Presence of severe hepatic disease or hepatic impairment
* Female who is pregnant or lactating
* Female of child-bearing potential not using adequate contraceptive measures
* Sexually active man with a partner of child-bearing potential who is not using adequate contraceptive measures
* Use of any prior and concomitant therapy which may interfere with the objective of the study
* Extensive tattoos

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients achieving T-VASI 50 on the body | From baseline to Day 140
  Measured using Vitiligo Area Scoring Index (VASI). A decrease in VASI indicates a reduction of the body surface area affected by vitiligo (possible range 1-100).

SECONDARY OUTCOMES:
Time to onset of repigmentation of full body | From baseline to first documented occurrence of TVASI25, assessed up to Day 140
  Measured using T-VASI 25. A decrease in VASI indicates a reduction of the total body surface area affected by vitiligo (possible range 1-100)
Time to onset of repigmentation of face | From baseline to first documented occurrence of FVASI25, assessed up to Day 140
  Measured using F-VASI 25. A decrease in VASI indicates a reduction of the total body surface area affected by vitiligo (possible range 1-100).
Percentage of patients achieving VASI 50 on the face | From baseline to Day 140
  Measured using VASI. A decrease in VASI indicates a reduction of the body surface area affected by vitiligo (possible range 1-100).
Percentage of patients maintaining VASI 50 on body surface area excluding hands and feet | From Day 140 to 308
  Measured using VASI. A decrease in VASI indicates a reduction of the body surface area affected by vitiligo (possible range 1-100).
Percentage of patients maintaining VASI 50 on facial lesions | From Day 140 to 308
  Measured using VASI. A decrease in VASI indicates a reduction of the body surface area affected by vitiligo (possible range 1-100).
Percentage of patients achieving VASI 25/75/90 on the body | From baseline to Day 140
  Measured using VASI. A decrease in VASI indicates a reduction of the body surface area affected by vitiligo (possible range 1-100).
Percentage of patients achieving VASI 25/75/90 on the face | From baseline to Day 140
  Measured using VASI. A decrease in VASI indicates a reduction of the body surface area affected by vitiligo (possible range 1-100).
Percentage change in pigmentation on body surface area measured by the VASI scoring system | From baseline to Day 308
  Measured using VASI. A decrease in VASI indicates a reduction of the body surface area affected by vitiligo (possible range 1-100).
Percentage change in pigmentation on facial surface area measured by the VASI scoring system | From baseline to Day 308
  Measured using VASI. A decrease in VASI indicates a reduction of the body surface area affected by vitiligo (possible range 1-100).

CONTACTS AND LOCATIONS:
Locations (30):
- United States (25):
  - CLINUVEL site, Birmingham, Alabama
  - CLINUVEL site, Fresno, California
  - CLINUVEL site, Los Angeles, California
  - CLINUVEL site, Palo Alto, California
  - CLINUVEL site, San Diego, California
  - CLINUVEL Site, Washington D.C., District of Columbia
  - CLINUVEL site, Miami, Florida
  - CLINUVEL site, Miramar, Florida
  - CLINUVEL site, Alpharetta, Georgia
  - CLINUVEL site, Augusta, Georgia
  - CLINUVEL site, Chicago, Illinois
  - CLINUVEL site, Baton Rouge, Louisiana
  - CLINUVEL site, Detroit, Michigan
  - CLINUVEL site, Minneapolis, Minnesota
  - CLINUVEL site, Roseville, Minnesota
  - CLINUVEL Site, Lee's Summit, Missouri
  - CLINUVEL site, Rochester, New York
  - CLINUVEL site, Cleveland, Ohio
  - CLINUVEL site, Philadelphia, Pennsylvania
  - CLINUVEL Site, Charleston, South Carolina
  - CLINUVEL site, Thompson's Station, Tennessee
  - CLINUVEL Site, Cedar Park, Texas
  - CLINUVEL site, Dallas, Texas
  - CLINUVEL site, Tyler, Texas
  - CLINUVEL site, Charlottesville, Virginia
- France (2):
  - CLINUVEL site, La Réunion
  - CLINUVEL site, Nice
- CLINUVEL site, Nairobi, Kenya
- United Kingdom (2):
  - CLINUVEL site, London
  - CLINUVEL site, Manchester